CLINICAL TRIAL: NCT06572631
Title: Phase 1b Expansion Study of Multi-Antigen Specific CD8+ T Cells After Decitabine-enhanced Lymphodepletion: An Adoptive Cellular Therapy for Patients With Relapsed or Refractory AML or MDS Following an Allogeneic Hematopoietic Cell Transplantation From Matched HLA Donors
Brief Title: Multi-antigen Specific CD8+ T Cells With Decitabine and Lymphodepleting Chemotherapy for the Treatment of Patients With Relapsed or Refractory AML or MDS Following an Allogeneic Hematopoietic Cell Transplantation From a Matched Donor
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: cprmc withdrawn
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23606; NCI-2024-06709 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23606 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Acute Myeloid Leukemia; Recurrent Myelodysplastic Syndrome; Refractory Acute Myeloid Leukemia; Refractory Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Specimen Handling; Biopsy; Cyclophosphamide; Decitabine; Injections; fludarabine; Leukapheresis; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (NEXI-001, decitabine, chemotherapy) (Experimental): DONOR: Donors undergo leukapheresis on study.
  PATIENTS: Patients may receive bridging therapy per standard of care ≥ 14 days prior to the start of cycle 1. Patients receive decitabine IV over 1 hour QD on day -3, -5 or -10 to day -1, lymphodepletion chemotherapy with fludarabine IV over 30 minutes QD and cyclophosphamide IV over 60 minutes QD on day -5 to -3 and then receive NEXI-001 IV over 30 minutes QD on days 1, 8 and 15 of cycle 1. Cycles repeat every 33 or 38 days in the absence of disease progression or unacceptable toxicity. If NEXI-001 cells remain and treatment criteria are met, patients may receive and additional cycle of decitabine IV over 1 hour QD on day -5 to -1 and NEXI-001 IV QD on days 1, 8 and 15 in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO during screening, bone marrow aspirate and/or bone marrow biopsy, PET/ CT scan or MRI and blood sample collection throughout the study.
  Interventions: Biological: Allogeneic CD8+ Leukemia-associated Antigens Specific T Cells NEXI-001; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Decitabine; Procedure: Echocardiography; Drug: Fludarabine; Procedure: Leukapheresis; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: Allogeneic CD8+ Leukemia-associated Antigens Specific T Cells NEXI-001 — Given IV
  Other Names: NEXI 001; NEXI-001; NEXI001
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase I trial tests the safety, side effects and best dose of NEXI-001 when given with decitabine and lymphodepleting chemotherapy in treating patients with acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory) following an allogeneic hematopoietic cell transplantation from a matched donor. NEXI-001 is a type of chimeric antigen receptor T cell therapy in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein on the patient's cancer cells is added to the T cells in the laboratory. The special receptor is called a chimeric antigen receptor (CAR). Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. Decitabine is in a class of medications called hypomethylation agents. It works by helping the bone marrow produce normal blood cells and by killing abnormal cells in the bone marrow. Lymphodepleting chemotherapy, with fludarabine and cyclophosphamide, helps kill cancer cells in the body and helps prepare the body for the new CAR-T cells. Giving NEXI-001 with decitabine and lymphodepleting chemotherapy may be safe and tolerable in treating patients with relapsed or refractory AML or MDS following an allogeneic hematopoietic cell transplantation from a matched donor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Characterize the safety of allogeneic CD8+ leukemia-associated antigens specific T cells NEXI-001 (NEXI-001) combined with decitabine.

II. Determine the recommended phase 2 dose (RP2D) for NEXI-001 T cells combined with decitabine.

SECONDARY OBJECTIVES:

I. Investigate the preliminary anti-leukemic activity of NEXI-001 T cells combined with decitabine based on:

Ia. Complete response (CR) rate; Ib. Overall response rate (ORR); Ic. Median duration of response; Id. 1-year overall survival (OS); Ie. 1-year progression-free survival (PFS). II. Cumulative incidence of acute graft-versus-host disease (aGVHD) of grades 2-4 and 3-4 at day 100 post first infusion of NEXI-001.

III. Cumulative incidence of chronic graft-versus-host disease (cGVHD) of all grades at 1 year post first infusion of NEXI-001.

IV. Characterize the T cells in the NEXI-001 product by immunophenotype and tumor antigen specificity.

V. Characterize NEXI-001 T cells in peripheral blood (PB) and bone marrow (BM) by immunophenotype and tumor antigen specificity.

VI. Expansion and persistence of NEXI-001 T cells in PB and BM.

EXPLORATORY OBJECTIVES:

I. Evaluate the effect of the following factors on the safety and efficacy of NEXI-001 T cells combined with decitabine:

Ia. NEXI-001 T-cell immunophenotype; Ib. Persistence of NEXI-001 T cells in PB and BM; Ic. Blood levels of the antigen-specific NEXI-001 T cells; Id. Biomarkers of activation, proliferation, and exhaustion of T cells; Ie. The expression of tumor associated antigen (TAAs) and checkpoint molecules on AML blasts.

OUTLINE: This is a dose-escalation study of decitabine in combination with NEXI-001, fludarabine and cyclophosphamide.

DONOR: Donors undergo leukapheresis on study.

PATIENTS: Patients may receive bridging therapy per standard of care ≥ 14 days prior to the start of cycle 1. Patients receive decitabine intravenously (IV) over 1 hour once per day (QD) on day -3, -5 or -10 to day -1, lymphodepletion chemotherapy with fludarabine IV over 30 minutes QD and cyclophosphamide IV over 60 minutes QD on day -5 to -3 and then receive NEXI-001 IV over 30 minutes QD on days 1, 8 and 15 of cycle 1. Cycles repeat every 33 or 38 days in the absence of disease progression or unacceptable toxicity. If NEXI-001 cells remain and treatment criteria are met, patients may receive and additional cycle of decitabine IV over 1 hour QD on day -5 to -1 and NEXI-001 IV QD on days 1, 8 and 15 in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography (ECHO) during screening, bone marrow aspirate and/or bone marrow biopsy, positron emission tomography (PET)/computed tomography (CT) scan or magnetic resonance imaging (MRI) and blood sample collection throughout the study.

After completion of study treatment, patients are followed up within 30 days and every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* PARTICIPANT: Documented informed consent of the participant and/or legally authorized representative and documented informed consent of the donor
* PARTICIPANT: Agreement to allow the use of archival tissue from diagnostic tumor biopsies (if unavailable, exceptions may be granted with study principal investigator [PI] approval)
* PARTICIPANT: Age: ≥ 18 years
* PARTICIPANT: Eastern Cooperative Oncology Group (ECOG) ≤ 1 or Karnofsky performance score (KPS) ≥ 70
* PARTICIPANT: Confirmed diagnosis of AML/MDS that has relapsed after or is refractory to an allogeneic hematopoietic cell transplantation (HCT) from a matched donor.

  * Refractory - failure to achieve a complete response minimal residual disease (CRMRD) (-) by multicolor flow cytometry (MFC) or reverse transcription polymerase chain reaction (RT qPCR)
  * Relapse - detection of clonal abnormal myeloid blasts by morphology (morphologic relapse) or by MFC, or RT-qPCR analysis (MRD[+] relapse) after achieving a CRMRD(-) induced by an allogeneic HCT or maintained by allogeneic HCT administered as consolidation therapy.

Note: Patients who meet the protocol definition of relapse/refractory (r/r) AML/MDS at screening and subsequently achieve a CRMRD(-) response status following protocol-specified bridging therapy will remain eligible to continue participation in this study

* PARTICIPANT: At least 100 days post allogeneic HCT
* PARTICIPANT: Donor match at 8 out of 8 loci for human leucocyte antigen (HLA) -A, -B, -C, and -DRB1 (each typed at high resolution by deoxyribonucleic acid [DNA]-based methods)
* PARTICIPANT: Expression of HLA-A*0201 as determined by high resolution sequence-based typing methods
* PARTICIPANT: Total bilirubin ≤ 1.5 X upper limit of normal (ULN) (unless has Gilbert's disease) (to be performed within 28 days of consenting)
* PARTICIPANT: Aspartate aminotransferase (AST) ≤ 2.5 x ULN (to be performed within 28 days of consenting)
* PARTICIPANT: Alanine aminotransferase (ALT) ≤ 2.5 x ULN (to be performed within 28 days of consenting)
* PARTICIPANT: Serum creatinine < 1.5 mg/dL or creatinine clearance of ≥ 60 mL/min per 24 hour urine test or the Cockcroft-Gault formula (to be performed within 28 days of consenting)
* PARTICIPANT: Left ventricular ejection fraction (LVEF) ≥ 50% Note: To be performed before the first dose of lymphodepletion chemotherapy
* PARTICIPANT: If able to perform pulmonary function tests: Forced expiratory volume in one second (FEV1), forced vital capacity (FVC), and diffuse lung capacity for carbon monoxide (DLCO) (diffusion capacity) ≥ 50% of predicted (corrected for hemoglobin) (to be performed within 28 days of consenting)
* PARTICIPANT: If unable to perform pulmonary function tests: Oxygen (O2) saturation > 92% on room air (to be performed within 28 days of consenting)
* PARTICIPANT: Seronegative for HIV antigen/antibody (Ag/Ab) combo, hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative), and syphilis (rapid plasma reagin [RPR]) (to be performed within 28 days of consenting)

  * If positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed. OR
  * If seropositive for HIV, HCV or HBV, nucleic acid quantitation must be performed. Viral load must be undetectable
* PARTICIPANT: Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required (to be performed within 28 days of consenting)
* PARTICIPANT: Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the completion of the last cycle of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* DONOR: The identified donor must be the donor whose stem cells were used for the research participant's allo HCT
* DONOR: The donor's hematocrit value is ≥ 35%
* DONOR: The donor's platelet count is > 100,000 per microliter
* CRITERIA TO PROCEED TO START OF CYCLE 1: NEXI-001 product is released from manufacturing with a certificate of analysis (COA)
* CRITERIA TO PROCEED TO START OF CYCLE 1: Bone marrow aspirate and bone marrow biopsy within one week prior to treatment for baseline disease status (all disease statuses are eligible to proceed) and correlative studies
* CRITERIA TO PROCEED TO START OF CYCLE 1: T-cell chimerism ≥ 50% to donor by polymerase chain reaction (PCR) analysis
* CRITERIA TO PROCEED TO START OF CYCLE 1: Fully recovered to ≤ grade 1 from non-hematologic acute toxic effects (except alopecia) from prior anti-cancer therapy
* CRITERIA TO PROCEED TO START OF CYCLE 1: Total bilirubin ≤ 1.5 X ULN (unless has Gilbert's disease) (to be performed within 2 days prior to start of cycle therapy)
* CRITERIA TO PROCEED TO START OF CYCLE 1: AST =< 2.5 x ULN (to be performed within 2 days prior to start of cycle therapy)
* CRITERIA TO PROCEED TO START OF CYCLE 1: ALT =< 2.5 x ULN (to be performed within 2 days prior to start of cycle therapy)
* CRITERIA TO PROCEED TO START OF CYCLE 1: Serum creatinine < 1.5 mg/dL or creatinine clearance of ≥ 60 mL/min per 24 hour urine test or the Cockcroft-Gault formula (to be performed within 2 days prior to start of cycle therapy)
* CRITERIA TO PROCEED TO START OF CYCLE 1: If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin (PT) ≤ 1.5 x ULN. If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants (to be performed within 2 days prior to start of cycle therapy)
* CRITERIA TO PROCEED TO START OF CYCLE 1: If not receiving anticoagulants: Activated partial thromboplastin Time (aPTT) ≤ 1.5 x ULN. If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants (to be performed within 2 days prior to start of cycle therapy)
* CRITERIA TO PROCEED TO START OF CYCLE 1: Left ventricular ejection fraction (LVEF) ≥ 50% (to be performed within 2 days prior to start of cycle therapy)

  * Note: To be performed before the first dose of LD chemotherapy
* CRITERIA TO PROCEED TO START OF CYCLE 1: Corrected QT (QTc) ≤ 480 ms (to be performed within 2 days prior to start of cycle therapy)
* CRITERIA TO PROCEED TO START OF CYCLE 1: O2 saturation > 92% on room air (to be performed within 2 days prior to start of cycle therapy)
* CRITERIA TO PROCEED TO START OF CYCLE 1: Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required (to be performed within 2 days prior to start of cycle therapy)
* CRITERIA TO PROCEED TO START OF CYCLE 1: Investigational drugs or devices within 30 days prior to start of cycle 1 therapy
* NEXI-001 INCLUSION CRITERIA: Total bilirubin ≤ 2.5 X ULN (unless has Gilbert's disease) (to be performed within 1 days prior to NEXI-001 infusion)
* NEXI-001 INCLUSION CRITERIA: AST =< 3 x ULN (to be performed within 1 days prior to NEXI-001 infusion)
* NEXI-001 INCLUSION CRITERIA: Serum creatinine < 2 mg/dL (to be performed within 1 days prior to NEXI-001 infusion)
* NEXI-001 INCLUSION CRITERIA: O2 saturation > 92% on room air (to be performed within 1 days prior to NEXI-001 infusion)
* CRITERIA TO PROCEED TO CYCLE 2: Patient has achieved a response of at least stable disease
* CRITERIA TO PROCEED TO CYCLE 2: ANC must be at least 1,000/uL and platelets at least 50,000/uL to begin decitabine
* CRITERIA TO PROCEED TO CYCLE 2: Patient has not experienced a ≥ grade 3 NEXI-001-related nonhematological AE that did not resolve to ≤ grade 2 within 72 hours

Exclusion Criteria:

* PARTICIPANT: Patients who have had 2 prior allogeneic (allo) HCTs
* PARTICIPANT: Patients who have received more than 3 anti-leukemic treatments regimens since their allo HCT
* PARTICIPANT: Vaccination with a live virus within six months prior to study treatment.

  * Inactivated influenza vaccination is allowed
* PARTICIPANT: Active acute or chronic GVHD
* PARTICIPANT: Known hypersensitivity to any component of the NEXI-001 T-cell product or fludarabine, cyclophosphamide, decitabine, or tocilizumab
* PARTICIPANT: Clinically significant uncontrolled illness
* PARTICIPANT: A second primary malignancy that has not been in remission for > 2 years. Exceptions include the following resected lesions:

  * Non-melanoma skin cancer.
  * Carcinoma in situ.
  * Squamous intraepithelial lesions on Pap smear.
  * Localized prostate cancer (Gleason score < 6).
  * Melanoma in situ
* PARTICIPANT: Females only: Pregnant or breastfeeding
* PARTICIPANT: Clinically significant cardiovascular disease:

  * Myocardial infarction or unstable angina within 6 months prior to the start of lymphodepleting (LD) chemotherapy.
  * Cerebral vascular accident or a transient ischemic attack within 6 months prior to the start of LD chemotherapy.
  * Clinically significant cardiac arrhythmia
  * Uncontrolled hypertension
  * Congestive heart failure (New York Heart Association Class III or IV)
  * Pericarditis or clinically significant pericardial effusion
  * Myocarditis
* PARTICIPANT: History of autoimmune disease resulting in end organ injury or requiring systemic immunosuppression or systemic disease modifying therapy within 2 years prior to enrollment.

  * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone remain eligible.
  * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen remain eligible
* PARTICIPANT: Major trauma or major surgery within 4 weeks of enrollment
* PARTICIPANT: Dementia or altered mental status that precludes understanding the informed consent form
* PARTICIPANT: History of seizures or other chronic clinically significant neurologic disorders.

  * Patients with well-controlled seizures on anti-seizure medication without a seizure episode for ≥ 6 months remain eligible
* PARTICIPANT: Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* PARTICIPANT: Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)
* DONOR: The donor is pregnant or breastfeeding at the time of requested donation
* DONOR: The donor had granulocyte colony stimulating factor (G-CSF) administered within one month, prior to leukapheresis
* DONOR: The donor has an active bacterial or fungal infection, which is currently not responding to antimicrobial treatment
* CRITERIA TO PROCEED TO START OF CYCLE 1: Other anti-leukemic (bridging) therapies within 14 days of start of cycle 1 therapy
* CRITERIA TO PROCEED TO START OF CYCLE 1: Patients receiving systemic corticosteroid (> 20 mg/day prednisone equivalent) or any other immunosuppressant agents at the time of initiation of LD chemotherapy. Intermittent topical, inhaled, or intranasal corticosteroids are allowed
* CRITERIA TO PROCEED TO START OF CYCLE 1: Active acute or chronic GVHD (Note: must have resolved by the time of initiation of cycle 1 of therapy
* CRITERIA TO PROCEED TO START OF CYCLE 1: Active or uncontrolled infection requiring antibiotics by the time LD chemotherapy is scheduled. Prophylactic and ongoing therapy for prior controlled infection is allowed
* CRITERIA TO PROCEED TO START OF CYCLE 1: Females only: Pregnant or breastfeeding
* CRITERIA TO PROCEED TO START OF CYCLE 1: Clinically significant cardiovascular disease:

  * Myocardial infarction or unstable angina within 6 months prior to the start of LD chemotherapy
  * Cerebral vascular accident or a transient ischemic attack within 6 months prior to the start of LD chemotherapy
  * Clinically significant cardiac arrhythmia
  * Uncontrolled hypertension
  * Congestive heart failure (New York Heart Association Class III or IV)
  * Pericarditis or clinically significant pericardial effusion
  * Myocarditis
  * History of seizures or other chronic clinically significant neurologic disorders. Patients with well-controlled seizures on anti-seizure medication without a seizure episode for ≥ 6 months remain eligible
* CRITERIA TO PROCEED TO START OF CYCLE 1: Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* NEXI-001 EXCLUSION CRITERIA: Patient has no evidence of NEXI-001-related nonhematological adverse events (AEs), e.g. cytokine release syndrome (CRS), immune effector cell-associated neurotoxicity syndrome (ICANS), hemophagocytic lymphohistiocytosis (HLH)/macrophage activation syndrome (MAS)
* NEXI-001 EXCLUSION CRITERIA: Patient has not developed any of the exclusion criteria for treatment
* CRITERIA TO PROCEED TO CYCLE 2: Patient has not developed any of the exclusion criteria for treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-07 (Estimated); Primary Completion 2026-12-12 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 1.5 years
  AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0, with the following exceptions: cytokine Release Syndrome will be graded according to the consensus criteria published by the American Society for Transplantation and Cellular Therapy, Immune effector Cell-Associated Neurotoxicity Syndrome, acute graft versus host disease (GVHD) grading according to Magic Consortium criteria and chronic GVHD grading according to National Health Institute Consensus criteria.
Dose limiting toxicity | Up to completion of cycle 1
  Defined as grade 3 or higher non-hematological AE excluding toxicities unequivocally related to underlying disease, intercurrent illness or alternative etiology, and with the following exceptions: grade 3 or higher cytokine release syndrome/neurotoxicity that responds to appropriate medical intervention within 72 hours before improving to < grade 2 and grade 3-4 GVHD if responsive to therapy within 14-21 days.

SECONDARY OUTCOMES:
Overall response | Up to 1.5 years
  By the 2022 European Leukemia Net criteria for acute myeloid leukemia (AML)/myelodysplastic syndrome (MDS). Will be analyzed using the Kaplan-Meier method.
Complete response | Up to 1.5 years
  By morphologic, multiparametric flow cytometry, and real time quantitative polymerase chain reaction criteria. Will be analyzed using the Kaplan-Meier method.
Duration of response | From the starting date of response to the date of disease progression, up to 1.5 years
  Will be analyzed using the Kaplan-Meier method.
Progression free survival | From starting study therapy to the first observation of disease progression or date of death, whichever comes first, up to 1.5 years
  Will be analyzed using the Kaplan-Meier method.
Overall survival | From starting study therapy to the date of death, up to 1.5 years
  Will be analyzed using the Kaplan-Meier method.
Determine the immunophenotype of NEXI-001 T cells | Up to 1.5 years
  In peripheral blood (PB) and bone marrow (BM) by flow cytometry techniques.
Incidence of acute GVHD | Up to 1.5 years
  Of grades 2-4 and 3-4 (grading according to Magic Consortium criteria). Will be calculated using death and disease progression as competing risks.
Incidence of chronic GVHD | Up to 1.5 years
  Of all grades (grading according to Lee et al. 2017). Will be calculated using death and disease progression as competing risks.
Persistence/antigen specificity of NEXI-001 T cells | Up to 1.5 years
  In PB and BM by multimer-based staining over time.

CONTACTS AND LOCATIONS:
Overall Officials: Monzr M Al Malki, MD, Principal Investigator — City of Hope Medical Center